CLINICAL TRIAL: NCT02227355
Title: A Multi-center Noninterventional Study to Evaluate the Effectiveness of Neupro® (Rotigotine Transdermal Patch) and Levodopa Combination Therapy in Patients With Parkinson's Disease (NEUPART)
Brief Title: Evaluating the Effectiveness of Neupro® (Rotigotine) and L-dopa Combination Therapy in Patients With Parkinson's Disease
Acronym: NEUPART
Status: Completed | Type: Observational
Sponsor: UCB Biopharma S.P.R.L. (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Other Study IDs: PD0013
Record Dates: First submitted 2014-08-26; First posted 2014-08-28 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-07

CONDITIONS: Idiopathic Parkinson's Disease
Keywords: Parkinson's Disease; Neupro®; Rotigotine; Transdermal patch; NEUPART; Levodopa; Noninterventional; Combination therapy
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PD Patients < 70 years of age: Patients with Parkinson's Disease (PD) <70 years of age.
- PD Patients ≥ 70 years of age: Patients with Parkinson's Disease (PD) ≥ 70 years of age.

SUMMARY:
This study aims to evaluate the effectiveness of Rotigotine and Levodopa combination therapy for younger and older patients with Parkinson's Disease under real life conditions. Effects on ability to perform activities of daily living, sleep, medication dose and other factors will be assessed.

ELIGIBILITY:
Inclusion Criteria:

The following selection criteria must be followed for patients entering the Noninterventional Study (NIS):

* The decision by the treating physician to prescribe Rotigotine transdermal patch is made before participating in the NIS due to a clinical therapeutic indication (e.g., because of intolerance and/or ineffectiveness of another dopamine agonist)
* The patient is either male or female and over 18 years of age
* A Patient Data Consent form is signed and dated by the patient or by the legal representative
* The patient has idiopathic Parkinson's Disease, has not received Rotigotine within 28 days prior to the Baseline Visit and is willing to participate in questionnaire based assessments
* The patient is receiving L-dopa as monotherapy or a combination therapy composed of L-dopa and a dopamine agonist other than Rotigotine
* The patient has been on L-dopa therapy for at least 6 months and is responding to initial L-dopa therapy
* The patient has a Hoehn and Yahr stage score of 1 to 4.

Exclusion Criteria:

* Patients will be excluded from the study if they have participated in a clinical study of a medication or a medical device within 3 months prior to Baseline or if they are participating in a clinical study at the time of inclusion or have already participated in the current study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with idiopathic Parkinson's Disease receiving levodopa as monotherapy or in combination with a dopamine agonist other than Rotigotine, but either not sufficiently controlled on or intolerant to current treatment, or other reason; patients are receiving treatment in general practitioner (GP) offices, private clinics or hospitals (including university hospitals) according to routine daily practice.
Sampling Method: Probability Sample
Enrollment: 195 (Actual)
Dates: Start 2014-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to end of the Observational Period in Unified Parkinson's Disease Rating Scale Part II (UPDRS Part II) total score | Baseline to end of Observational Period (6 months)
  The UPDRS Part II (Activities of Daily Living) consists of 13 items, each to be scored between 0 (normal/none) and 4 (highest level of severity). The sum score is calculated as the sum of the 13 individual scores (13 questions=52 points maximum; the higher the sum score, the greater degree of disability).

SECONDARY OUTCOMES:
Change from Baseline to end of the Observational Period in L-dopa dose | Baseline to end of Observational Period (6 months)
Change from Baseline to end of the Observation Period in Parkinson's Disease Sleep Scale (PDSS-2) total score | Baseline to end of Observational Period (6 months)
  The PDSS-2 is a 15 item scale that is used to assess sleep and nocturnal disability in Parkinson's Disease. It is designed for interviewer-administered completion or self-completion by patients.
  Patients are asked to rate how often during the past week he/she slept well or experienced various symptoms of sleep disability. Each of the 15 items are to be scored between 0 (never) to 4 (very often) with the total score ranging from 0 to 60; the higher the sum score, the greater the degree of impairment.
Response at the end of the Observation Period defined as 20 % decrease in Unified Parkinson's Disease Rating Scale Part II (UPDRS Part II) total score | End of the Observation Period (Month 6)
  The UPDRS Part II (Activities of Daily Living) consists of 13 items, each to be scored between 0 (normal/none) and 4 (highest level of severity). The sum score is calculated as the sum of the 13 individual scores (13 questions = 52 points maximum); the higher the sum score, the greater degree of disability.
Assessment at the end of the Observation Period in the score of the Clinical Global Impressions (CGI) Item 2 (Global Rating of Change of Condition) | End of the Observation Period (Month 6)
  CGI Item 2 (Global Rating of Change of Condition) requires the clinician to rate how much the patient's illness has improved or worsened relative to a baseline state. Scores range from 0 to 7 as follows: 0=not assessed, 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, 7=very much worse.

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (42):
- France (3):
  - 42, Lille
  - 41, Mougins
  - 40, Nîmes
- Germany (15):
  - 6, Alzenau in Unterfranken
  - 51, Aschaffenburg
  - 13, Beelitz-Heilstätten
  - 12, Berlin
  - 5, Böblingen
  - 53, Düsseldorf
  - 7, Erbach im Odenwald
  - 4, Haag
  - 11, Leer
  - 2, Münster
  - 54, Schriesheim
  - 8, Senftenberg
  - 14, Tübingen
  - 10, Ulm
  - 3, Westerstede
- Italy (9):
  - 45, Ancona
  - 47, Brescia
  - 60, Cagliari
  - 29, Cosenza
  - 30, Florence
  - 46, Milan
  - 27, Napoli
  - 28, Roma
  - 62, Roma
- Spain (4):
  - 20, Barakaldo
  - 15, Donostia / San Sebastian
  - 24, Madrid
  - 22, Palma de Mallorca
- United Kingdom (11):
  - 37, Bury
  - 49, Cambridge
  - 52, Lincoln
  - 48, Liverpool
  - 33, London
  - 36, London
  - 34, Manchester
  - 31, Middlesbrough
  - 38, North Shields
  - 35, Norwich
  - 63, Plymouth